CLINICAL TRIAL: NCT06406192
Title: Effects of Facilitating On-Site Recordings of Office Blood Pressure, Height, and Weight on Preventive Medicine - A Pragmatic Cluster Randomized Trial
Brief Title: Effects of FOR-Care Model on Preventive Medicine
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202402048RIND
Record Dates: First submitted 2024-04-28; First posted 2024-05-09 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus; Body Weight; Family Medicine; Hypertension; Preventive Medicine
Keywords: Body weight; Diabetes mellitus; Cluster randomized trial; Family medicine; Outpatient department; Preventive medicine
MeSH Terms: conditions — Diabetes Mellitus; Body Weight; Hypertension | interventions — Body Height

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No Intervention Group (No Intervention): This group does not specifically encourage or interfere with physicians' original methods of inquiry or patients providing bodily examination data.
- Intervention Group (Experimental): This group encourages physicians to actively inquire or patients to voluntarily provide physical examination data during consultations.
  Interventions: Diagnostic Test: Height, Weight, and Blood Pressure Measurement Procedures Improvement

INTERVENTIONS:
Diagnostic Test: Height, Weight, and Blood Pressure Measurement Procedures Improvement — In the intervention group, the investigators improve the process of measuring blood pressure, height, and weight, requiring timely recording of these measurements. The intervention includes:
  i. Enlisting the assistance of nurses and volunteers to improve the accessibility of measurement environments and provide guidance on instrument operation.
  ii. Using paper reminders at check-in stations to prompt patients to complete blood pressure and weight recordings before entering examination rooms; providing paper for recording if patients forget their health insurance cards.
  iii. Providing alcohol and hand wipes outside examination rooms for disinfecting measurement instruments.
  iv. Promoting the recording mode outside the check-in station.
  v. Ensuring that physicians or nurses in examination rooms accurately record measurements in the medical order system.
  vi. Encouraging patients to ask physicians during consultations, "Is my blood pressure and weight okay?"
  Other Names: FOR-Care Model
  Arms: Intervention Group

SUMMARY:
This study aims to address the prevalence of undiagnosed hypertension and diabetes by assessing the impact of the FOR-Care model on preventive medicine. The model focuses on improving the documentation of blood pressure, height, and weight in outpatient settings. Through a cluster randomized trial at National Taiwan University Hospital, clinics will either implement the FOR-Care model or continue with usual care. The trial will evaluate the effectiveness of the intervention in documenting these measurements and its impact on diagnosing hypertension and diabetes. The outcomes will provide valuable insights into enhancing preventive medicine and improving care for chronic diseases.

DETAILED DESCRIPTION:
Background: The prevalence of undiagnosed hypertension and diabetes among adults is considerable. For those already diagnosed with hypertension and diabetes, monitoring blood pressure and controlling body weight are recognized as essential methods for risk assessment. However, in outpatient settings, there is still room for improvement in the on-site documentation of blood pressure, height, and weight.

Objective: This cluster randomized trial (CRT) will assess the effects of preventive medicine following the implementation of the FOR-Care model, a technique designed for facilitating on-site recordings of office blood pressure, height, and weight.

Methods: The investigators will conduct a pragmatic CRT at the outpatient clinics of the Department of Family Medicine, National Taiwan University Hospital. A total of 42 clinics with over 15 patients will be randomized into two groups. The intervention group will adopt a FOR-Care model, required to measure and record blood pressure, height, and weight before consultations; while the control group receives usual care. The protected medical information will be accessed through the National Taiwan University Hospital Integrative Medical Database (NTUH-iMD). The quality improvement outcome is documentation of on-site blood pressure, height, and weight recordings of both groups at 12 and 24 weeks (cluster-level parameter). The primary preventive medicine outcome is newly diagnosed hypertension and diabetes mellitus (individual-level parameter). The secondary preventive medicine outcomes are clinical indicators of hypertension and diabetes mellitus in those with these diagnoses (individual-level parameters).

Expected Outcomes: The results of this pragmatic CRT will shed new insight into preventive medicine and quality of care in the management of common chronic diseases.

ELIGIBILITY:
Cluster-level inclusion criteria:

* clinic sessions with at least 15 patients, but fewer than 40 patients

Cluster-level exclusion criteria:

* travel, hospice, vaccination, or health examination clinics
* special-appointed clinics

Patient-level exclusion criteria

* patients aged less than 18
* patients with active catastrophic illness or terminal malignancies
* patients with major adverse cardiac events within 3 months before the index dates

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with Documented On-Site Blood Pressure, Height, and Weight Recordings | From enrollment to the next follow-up visit at either 12 weeks or 24 weeks afterward
  The documentation of on-site blood pressure, height, and weight recordings
Rate of Newly-Diagnosed Hypertension | From enrollment to the next follow-up visit at either 12 weeks or 24 weeks afterward
  Assessing whether the improvement in documentation of on-site blood pressure, height, and weight recordings increases the diagnosis rates of hypertension.
Rate of Newly-Diagnosed Diabetes Mellitus | From enrollment to the next follow-up visit at either 12 weeks or 24 weeks afterward
  Assessing whether the improvement in documentation of on-site blood pressure, height, and weight recordings increases the diagnosis rates of diabetes mellitus.

SECONDARY OUTCOMES:
Office Blood Pressure in Hypertensionsive Patients | From enrollment to the next follow-up visit at either 12 weeks or 24 weeks afterward
  Assessing whether the intervention affects clinical indicators of hypertension
Home Blood Pressure in Hypertensionsive Patients | From enrollment to the next follow-up visit at either 12 weeks or 24 weeks afterward
  Assessing whether the intervention affects clinical indicators of hypertension
Estimated Glomerular Filtration Rate | From enrollment to the next follow-up visit at either 12 weeks or 24 weeks afterward
  Assessing whether the intervention affects renal function (all patients)
Urinary Microalbumin Excretion | From enrollment to the next follow-up visit at either 12 weeks or 24 weeks afterward
  Assessing whether the intervention affects renal function (all patients)
Mortality Rate | From date of randomization until the date of first documented progression, assessed up to 36 months
  Assessing whether the intervention affects longterm survival status

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hsieh Chiang, MD, MPH, PhD, Study Chair — Family MedicineClinical Assistant Professor, Department of Family Medicine
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
However, de-identified data regarding the pre-defined outcomes or relevant characteristics could be available per request.